CLINICAL TRIAL: NCT03775330
Title: Parallel Prospective Observational Cohorts Evaluating Stereotactic Radiosurgery Alone (SRS) and Whole Brain Radiotherapy (WBRT) Plus SRS for Patients With 5 to 30 Brain Metastases
Brief Title: Radiosurgery With or Without Whole Brain Radiation for Multiple Metastases
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: BRAIN METS SRS
Record Dates: First submitted 2018-03-21; First posted 2018-12-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-09

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SRS: Stereotactic radiosurgery
  Interventions: Radiation: Stereotactic Radiosurgery (SRS)
- SRS plus WBRT: Stereotactic radiosurgery plus whole brain radiation
  Interventions: Radiation: Stereotactic Radiosurgery (SRS); Radiation: Whole brain radiation (WBRT)

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery (SRS) — SRS or hypofractionated stereotactic radiation delivered via the Leksell Gammknife Perfexion/Icon radiosurgery system. Hypofractionated stereotactic radiotherapy 25-32.5 Gy in 5 fractions or 24-27 Gy in 3 fractions at the discretion of the radiation oncologist
  Maximum diameter of metastasis (doses in single fraction):
  ≤ 2 cm: 15-20 Gy > 2 cm and ≤ 3 cm: 15-18 Gy > 3 cm and ≤ 4 cm: 15 Gy
  Tumour location (doses in single fraction):
  Brainstem: 15 Gy
  Hypofractionated stereotactic radiotherapy 25-32.5 Gy in 5 fractions may be used for lesions > 2 cm at the discretion of the radiation oncologist
  Note: SRS dosing reduced by 20% (for all prescriptions > 15 Gy) when patient is randomized to SRS + WBRT arm
Radiation: Whole brain radiation (WBRT) — WBRT 20 Gy in 5 fractions or 30 Gy in 10 fractions at the discretion of the radiation oncologist
  Groups: SRS plus WBRT

SUMMARY:
This clinical study is a parallel, prospective observational single-centre trial in patients presenting with 5 to 30 brain metastases. Patients to receive either stereotactic radiosurgery (SRS) alone or SRS plus whole brain radiation (WBRT) will be enrolled.

DETAILED DESCRIPTION:
The current standard of care for patients with limited brain metastases (1 to 4) is stereotactic radiosurgery (SRS) alone. This has evolved from the traditional standard of care in treating patients with whole brain radiation (WBRT). Studies in patients with limited (less than 5) brain metastases have shown that WBRT is harmful with respect to neurocognition and does not improve patient survival compared to SRS alone. As a result, SRS alone now is considered the standard of care treatment for patients with limited metastases. However, there is a lack of high quality prospective randomized evidence on the role of SRS in patients with 5 or more brain metastases to guide treatment.

Therefore, this study seeks to prospectively compare SRS alone versus SRS plus WBRT in patients with 5 to 30 brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of non-hematopoietic malignancy (excluding germ cell malignancies and small cell carcinoma).
* Patients with ≥ 5 but ≤ 30 de novo brain metastases seen on a diagnostic-quality contrast-enhanced MRI obtained within 30 days prior to enrollment (or randomization if previously randomized). Patients who are found to have 31-50 metastatic lesions at the time of treatment planning may still participate in the study. Disease progression such that > 50 brain metastases are detected after initial MRI prior to enrollment but before SRS will be treated off-protocol as per discretion of the treating physician.
* Patients with ≥ 5 but ≤ 30 new brain metastases who have undergone prior SRS for 4 or less brain metastases with stable intracranial disease as per diagnostic MRI for at least 6 months post last course of SRS. Patients who are found to have 31-50 new metastatic lesions at the time of treatment planning may still participate in the study. Disease progression such that > 50 new brain metastases are detected after initial MRI prior to enrollment but before SRS will be treated off-protocol as per discretion of the treating physician.
* Age ≥ 18.
* Karnofsky Performance Status (KPS) ≥ 70.
* Baseline HVLT-R above ≥ 6
* Patients must be able to tolerate WBRT, and all brain lesions must be eligible for treatment with SRS as determined by the radiation oncologist.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patient is able to read, speak, and understand (i.e. sufficiently fluent) English in order to allow completion and meaningful analyses of the neurocognitive tests and quality of life questionnaires.
* Patients must be accessible for treatment and follow up. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Patients who are on immunotherapy must have immunotherapy held at least 1 week before and after completion of radiotherapy. Other targeted agents/therapy must be held at least 1 day before and after SRS. Systemic chemotherapy must be held one week prior to treatment and re-started one week after treatment is complete.
* Protocol treatment is to begin within 4 weeks of patient enrollment (or randomization if previously randomized).

Exclusion Criteria:

* Patients with brain metastases resulting from germ cell malignancies, small cell carcinoma, or hematologic malignancies.
* Prior SRS for 5 or more brain metastases or any SRS for brain metastases within the last 6 months.
* Any prior WBRT or radiotherapy for brain metastases such that the study interventions cannot be delivered.
* Prior surgical resection of metastatic cancer from the brain.
* Patients with evidence of leptomeningeal disease.
* Patients who have a pacemaker or other contraindications, such that gadolinium-enhanced MRI cannot be performed or treatment cannot be delivered safely.
* Patients who have received chemotherapy or immunotherapy within 1 week prior to administration of protocol radiotherapy or who are expected / planned to receive chemotherapy within one week of completing protocol radiotherapy.
* Patients with < 5 or > 30 de novo or new brain metastases at time of enrollment, or > 50 brain metastases at time of treatment planning.
* Patients who are pregnant (women of child-bearing age must have negative pregnancy urine test within 7 days of enrollment or randomization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participant population will be patients who have MRI-documented 5 to 30, inclusive, brain metastases at time of enrollment and who are suitable for receiving stereotactic radiosurgery (SRS) and whole brain radiation (WBRT), with or without hippocampal-avoidance.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive function | 2 months post treatment
  Hopkins Verbal Learning Test-Revised (HVLT-R) Total Recall using the Reliable Change Index (RCI)

SECONDARY OUTCOMES:
Neurocognitive function - HVLT-R | 2 months, 4 months, 6 months, and 9 months
  Hopkins Verbal Learning Test-Revised (HVLT-R) (Total Recall, Delayed Recall, Delayed Recognition)
Neurocognitive function - Trail Making Test | 2 months, 4 months, 6 months, and 9 months
  Trail Making Test (TMT, Part A and Part B)
Neurocognitive function - Controlled Oral Word Association | 2 months, 4 months, 6 months, and 9 months
  Controlled Oral Word Association (COWA)
Neurocognitive function - Clinical Trial Battery Composite | 2 months, 4 months, 6 months, and 9 months
  Clinical Trial Battery Composite (CTB COMP) score
Local control of sites initially treated by SRS | 2 months, 4 months, 6 months, and 9 months
  Defined by the response criteria stipulated in the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria guideline
Distant tumour control within the brain | 2 months, 4 months, 6 months, and 9 months
  Distant brain failure is defined as the appearance of one or more new lesions on a diagnostic-quality, contrast-enhanced MRI within the brain at sites other than those initially treated by SRS
Overall central nervous system (CNS) response | 2 months, 4 months, 6 months, and 9 months
  Response will be recorded for each individual target lesion and for overall central nervous system (CNS) response as a composite of radiographical CNS target and non-target lesion responses, corticosteroid use, and clinical status defined as per RANO-BM criteria
Overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 36 months
  Response recorded for survival
Measure of Quality of Life | 2 months, 4 months, 6 months, and 9 months
  Health-Related QoL as measured by Functional Assessment of Cancer Therapy - Brain (FACT-Br) instrument
Incidence of Brain Salvage therapy During Follow-up | 2 months, 4 months, 6 months, and 9 months
  Number/proportion of patients requiring salvage therapy and type of salvage therapy, for progressive intracranial disease during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Lin Tseng, M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No